CLINICAL TRIAL: NCT01582997
Title: An Open-label, Dose Escalation, Phase I Study to Evaluate the Safety, Tolerability and Pharmacokinetic Profile of GSK2118436 in Japanese Subjects With BRAF V600 Mutation Positive Solid Tumors
Brief Title: A Phase I Study to Investigate the Safety, Tolerability and Pharmacokinetic Profile of of GSK2118436 in Japanese Subjects With BRAF Mutation Positive Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 116056
Record Dates: First submitted 2012-04-05; First posted 2012-04-23 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Cancer
Keywords: BRAF; Advance solid tumors
MeSH Terms: conditions — Neoplasms | interventions — dabrafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dose Escalation Part (Experimental): Dose escalation will be conducted to assess safety, tolerability, single and repeat dose PK profile and preliminary efficacy of GSK2118436 . The dose may be escalated to the overseas recommended phase III dose.
  Interventions: Drug: GSK2118436

INTERVENTIONS:
Drug: GSK2118436 — Dose escalation with GSK2118436 may proceed until the overseas recommended phase III dose.

SUMMARY:
BRF116056 is the first clinical experience with GSK2118436, a BRAF inhibitor, in Japan. This study will be designed to assess safety, tolerability, single and repeat dose PK profile and preliminary efficacy of GSK2118436 in Japanese subjects with BRAF V600 mutation positive solid tumors using continuous daily dosing schedule.

DETAILED DESCRIPTION:
BRF116056 is the first clinical experience with GSK2118436, a BRAF inhibitor, in Japan. This study will be designed to assess safety, tolerability, single and repeat dose PK profile and preliminary efficacy of GSK2118436 in Japanese subjects with BRAF V600 mutation positive solid tumors using continuous daily dosing schedule. Dose escalation of GSK2118436 will be performed according to a standard 3+3 dose-escalation design. GSK2118436 is given twice a day. However, to characterize the PK of GSK2118436 and its metabolites after single-dose administration, GSK2118436 will NOT be administrated for a week after the first administration. GSK2118436 continuous dosing will start after the 168-hour PK sample is obtained. Subjects may receive study treatment until disease progression, death or an unacceptable adverse event.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of a solid tumor that is not responsive to standard therapies or for which there is no approved or curative therapy.
* Subjects must have BRAF V600E or K mutant positive tumors.
* Women with reproductive potential must be willing to practice acceptable methods of birth control during the study and for up to 4 weeks after the last dose of study medication.
* Men with reproductive potential must be willing to practice acceptable methods of birth control during the study and for up to 16 weeks after the last dose of study medication.
* Must have adequate organ function.
* Must have Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1.

Exclusion Criteria:

* Currently receiving cancer therapy (chemotherapy, radiation therapy, immunotherapy, biologic therapy or surgery).
* Use of an investigational anti-cancer drug within 28 days preceding the first dose of GSK2118436.
* A history of other malignancy. Subjects who have been disease-free for 5 years or subjects with a history of complete resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible.
* History of Human Immunodeficiency Virus (HIV) infection.
* Certain cardiac abnormalities.
* Pregnant or lactating female.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-05-11 (Actual); Primary Completion 2014-08-01 (Actual); Study Completion 2015-04-16 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | First 28 days for Dose-limiting toxicity, Adverse Events for 1 year
  Adverse Events will be graded by the investigator according to the NCI-CTCAE (version 4.0)

SECONDARY OUTCOMES:
Pharmacokinetics (PK) parameters of GSK2118436 and its metabolites including blood concentration, Cmax and AUC | For 1 year
Tumor response as defined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | For 1 year
Serum levels of cytokines | For 1 year
Expression levels of pERK and Ki67 in tumor tissues if possible | For 1 year
Gene mutation in tumor tissues, including BRAF and KRAS | For 1 year

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Japan (2):
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokyo

REFERENCES:
- [Derived] Fujiwara Y, Yamazaki N, Kiyohara Y, Yoshikawa S, Yamamoto N, Tsutsumida A, Nokihara H, Namikawa K, Mukaiyama A, Zhang F, Tamura T. Safety, tolerability, and pharmacokinetic profile of dabrafenib in Japanese patients with BRAF V600 mutation-positive solid tumors: a phase 1 study. Invest New Drugs. 2018 Apr;36(2):259-268. doi: 10.1007/s10637-017-0502-8. Epub 2017 Sep 7. PMID 28879519
- See also: Results for study 116056 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/116056?search=study&search_terms=116056#rs